CLINICAL TRIAL: NCT00062036
Title: Tumor Infiltrating Lymphocytes (TIL Cells) Transduced With An Interleukin-2 (SBIL-2) Gene Following The Administration Of A Nonmyeloablative But Lymphocyte Depleting Regimen in Metastatic Melanoma
Brief Title: Cyclophosphamide and Fludarabine Followed By Interleukin-2 Gene-Modified Tumor Infiltrating Lymphocytes in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven A. Rosenberg, M.D./National Cancer Institute, National Institutes of Health
Masking: None | Purpose: Treatment
Other Study IDs: 030162; 03-C-0162; NCI-5855; CDR0000304438; NCT00059163 (obsolete NCT alias)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-03

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Filgrastim; incomplete Freund's adjuvant; Interleukin-2; Cyclophosphamide; fludarabine phosphate

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Biological: incomplete Freund's adjuvant
Biological: interleukin-2 gene
Biological: therapeutic tumor infiltrating lymphocytes
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as cyclophosphamide and fludarabine use different ways to stop tumor cells from dividing so they stop growing or die. Inserting the gene for interleukin-2 into a person's tumor infiltrating lymphocytes may make the body build an immune response to kill tumor cells. Combining cyclophosphamide and fludarabine with gene-modified tumor cells may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of gene-modified tumor infiltrating lymphocytes when given together with cyclophosphamide and fludarabine and to see how well they work in patients with metastatic melanoma (phase I is closed to accrual 3/29/06).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the survival of patients with metastatic melanoma administered interleukin-2 gene-modified tumor infiltrating lymphocytes after cyclophosphamide and fludarabine.
* Compare survival results with prior Surgery Branch studies using adoptive cell therapy without the interleukin-2 retroviral vector (SBIL-2) gene.

Secondary

* Determine clinical tumor regression in patients administered interleukin-2 gene-modified TIL after cyclophosphamide and fludarabine followed by interleukin-2.
* Determine the toxicity profile of this regimen in these patients.

OUTLINE:

* Phase I (closed to accrual as of 3/29/06):

  * Harvest: TIL are harvested, transduced with IL-2 gene, and expanded in vitro over a period of approximately 4 weeks.
  * Nonmyeloablative preparative regimen (chemotherapy): Patients receive cyclophosphamide IV over 1 hour on days -7 and -6 and fludarabine IV over 30 minutes on days -5 to -1.
  * Lymphocyte administration: Patients receive IL-2 gene-transduced TIL IV over 20-30 minutes on day 0. They also receive high-dose IL-2 IV over 15 minutes every 8 hours on days 0 -5 (maximum 15 doses). Beginning 1-2 days after lymphocyte administration, patients receive filgrastim (G-CSF) subcutaneously (SC) daily, , until blood counts recover.
  * Retreatment: Patients are re-evaluated every 4-6 weeks. Retreatment depends on disease status after each regimen. Patients with dose-limiting toxicity do not receive further treatment.

    * No response: Patients with stable disease or disease progression after the initial treatment are followed or removed from the study.
    * Partial response: Patients with a partial or minor response after the initial treatment may receive retreatment, approximately 2-4 weeks later, with chemotherapy, IL-2 gene-transduced TIL, immunization, and high-dose IL-2 as above, every 4-6 weeks for up to 2 courses provided at least a partial response is documented after each regimen.
    * Complete response: Patients with a complete response receive no further treatment.
* Phase II: Patients receive treatment and retreatment as in phase I with the MTD of IL-2 gene-transduced TIL.

Patients are followed every 3-6 weeks in the absence disease progression.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma

  * Metastatic disease
  * Refractory to standard therapy including high-dose interleukin-2 (IL-2) therapy
* Evaluable disease
* Patients may enroll at the cell infusion stage provided they have tumor available for biopsy OR expandable SBIL-2-transduced tumor infiltrating lymphocytes available
* Progressive disease during prior immunization to melanoma antigens or cellular therapy, with or without myeloablation, allowed
* Symptomatic CNS lesions allowed provided immediate active treatment for symptomatic lesions has been completed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count greater than 1,000/mm^3
* WBC greater than 3,000/mm^3
* Lymphocyte count greater than 500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 8.0 g/dL
* No coagulation disorder

Hepatic

* Bilirubin no greater than 2.0 mg/dL (less than 3.0 mg/dL in patients with Gilbert's syndrome)
* AST/ALT less than 3 times upper limit of normal
* Hepatitis B surface antigen negative
* Hepatitis C virus negative

Renal

* Creatinine no greater than 1.6 mg/dL

Cardiovascular

* No myocardial infarction
* No cardiac arrhythmias
* No abnormal stress thallium or comparable test
* LVEF > 45% and normal stress cardiac test in patients with the following criteria:

  * 50 years old or greater
  * History of EKG abnormalities, symptoms of cardiac ischemia or arrhythmias
* No major cardiovascular illness

Pulmonary

* No obstructive or restrictive pulmonary disease
* No major respiratory illness
* FEV_1 > 60% predicted in patients with prolonged history of cigarette smoking or symptoms of respiratory dysfunction

Immunologic

* HIV negative
* No prior severe immediate hypersensitivity reaction
* No primary or secondary immunodeficiency
* No active systemic infection
* No concurrent opportunistic infection
* No major immune system illness

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after study therapy
* Must sign a durable power of attorney

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior anti-cytotoxic T-lymphocyte antibody-4 antibody (CTLA-4) allowed unless post-MDX010 treatment and colonoscopy with colonic biopsies are normal

Chemotherapy

* Recovered from prior chemotherapy

Endocrine therapy

* No concurrent steroids

Radiotherapy

* Recovered from prior radiotherapy

Surgery

* Not specified

Other

* More than 4 weeks since prior systemic therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2003-06; Primary Completion 2007-02 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Clinical tumor regression
Toxicity profile

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland